CLINICAL TRIAL: NCT05415917
Title: Adjuvant Gemcitabine and Capecitabine Chemotherapy in Resected Pancreatic Cancer Following Neoadjuvant Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Prateek Gulhati, MD, PhD, Assistant Professor, Department of Gastrointestinal Medical Oncology, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CINJ 072206; Pro2022000669 (Other: Rutgers, The State University of New Jersey)
Record Dates: First submitted 2022-05-09; First posted 2022-06-13 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Pancreatic Cancer
Keywords: Gemcitabine Chemotherapy; Capecitabine Chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Capecitabine

STUDY DESIGN:
Intervention Model Description: A chemotherapy cycle will constitute 28 days of treatment:
  1. Gemcitabine: 1000 mg/m2 IV on days 1, 8, and 15 of each 28-day cycle
  2. Capecitabine: 1660 mg/m2 per day orally on days 1 through 21 of each 28-day cycle.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1- Gemcitabine and Capecitabine Treatment (Experimental): Day 1, Day 8, Day 15 • Gemcitabine infused through a vein over 120 minutes
  Day 1 - Day 21
  • Capecitabine tablets will be taken two times a day; once in the morning and once in the evening. The tablets should not be crushed or split and should be taken with a full glass of water (8 ounces/240 milliliters) within 30 minutes after a meal.
  Interventions: Drug: Gemcitabine and Capecitabine
- Group 2 - Observational (No Intervention): Usual therapy used to treat this type of cancer, chemotherapy plus radiation therapy. If cancer returns during observation, there will be offered standard of care therapy. Follow-up visits will be every three months.

INTERVENTIONS:
Drug: Gemcitabine and Capecitabine — A chemotherapy cycle will constitute 28 days of treatment:
  1. Gemcitabine: 1000 mg/m2 IV on days 1, 8, and 15 of each 28-day cycle
  2. Capecitabine: 1660 mg/m2 per day orally on days 1 through 21 of each 28-day cycle.
  Arms: Group 1- Gemcitabine and Capecitabine Treatment

SUMMARY:
Primary Objectives:

To determine the disease free survival (DFS) for participants treated with post-operative adjuvant chemotherapy, as compared to neoadjuvant therapy alone.

Secondary Objectives:

To determine the clinical efficacy of the study treatment in terms of median overall survival (OS) and median disease free survival (DFS).

To assess the safety and tolerability of the study treatment regimen as measured by the adverse events rates.

To assess the quality of life in patients receiving the study treatment.

DETAILED DESCRIPTION:
The purpose of the research is to compare the usual treatment approach (chemotherapy followed by surgery) to using chemotherapy followed by surgery and then more chemotherapy. This study will help the study doctors find out if this different approach is better, the same, or worse than the usual approach. To decide if it is better, the study doctors will be looking to see if the study approach increases the lifespan of patients compared to the usual approach. There will be two arms of the study. Arm one will receive treatment with gemcitabine and capecitabine every 28 days for 6 cycles. Arm two be will receive standard of care observation. Participants will be asked to undergo imaging (e.g., CT) and laboratory testing to monitor for disease recurrence. The time in the study will be for 30 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically confirmed diagnosis of pancreatic ductal adenocarcinoma
* Neoadjuvant chemotherapy (for at least three months) ± chemoradiation followed by R0 surgical resection
* Eastern Cooperative Oncology Group(ECOG) Performance status of PS 0 - 2
* At least 18 years of age
* Adequate bone marrow and organ functions as defined by:

  * Absolute neutrophil count ≥ 1000 cells/ μL
  * Hemoglobin ≥ 8 g/ dL
  * Platelets > 75,000 / μL
  * Creatinine ≤ 1.5 x ULN OR creatinine clearance ≥ 30 mL/min by Cockroft-Gault
  * Total bilirubin ≤1.5 ULN
  * AST/ ALT < 2.5 x ULN, unless with liver metastases and then must be <5 x ULN of normal
* Women and men of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect pregnancy on study, she must notify her treating physician immediately
* Ability to understand the nature of this study protocol and give written informed consent.
* Willingness and ability to comply with scheduled visits, treatment plans laboratory tests and other study procedures

Exclusion Criteria:

* Receipt of any investigational agents at the time of registration
* Known, untreated brain metastases
* Presence of metastatic disease or malignant ascites on diagnostic imaging
* Grade two or greater peripheral neuropathy
* Presence of any additional active malignancy within the past 3 years where the malignancy is at least reasonably likely to later the course of therapy, require systemic therapy or interfere with imaging assessments
* Uncontrolled intercurrent illness, including significant active infection, symptomatic congestive heart failure (NYHA classification grade III or IV), unstable angina or active arrhythmia
* Major surgery within the 4 weeks prior to initiation of study treatment
* A history of allergy or hypersensitivity to any of the study drugs
* Any additional significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from fully participating in the study
* Pregnancy
* Severe hepatic impairment
* Participants with known malabsorption

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by number of participants experiencing adverse events | Five Years
  Number of participants experiencing adverse events as defined by Cancer Therapy Evaluation Program Common Toxicity Criteria (CTC) Version 5.0 for toxicity

OTHER OUTCOMES:
To measure the tumor with the Response Evaluation Criteria in Solid Tumors (RECIST) | Five Years
  Response and progression will be evaluated in this study using the international criteria proposed by the revised Response Evaluation Criteria in Solid Tumors (RECIST) guidelines (version 1.1), when possible eleven Changes in the largest diameter (unidimensional measurement) of the tumor lesions and the shortest diameter in the case of malignant lymph nodes are used for tumor measurements. Imaging for response assessment will be obtained before the initiation of conditioning and at the six-week follow up time point.

CONTACTS AND LOCATIONS:
Overall Officials: Prateek Gulhati, MD, PhD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No